CLINICAL TRIAL: NCT00287508
Title: Emboshield and Xact Post Approval Carotid Stent Trial Using the Emboshield® BareWire™ Rapid Exchange Embolic Protection System and Xact® Rapid Exchange Carotid Stent System
Brief Title: Emboshield® and Xact® Post Approval Carotid Stent Trial (The EXACT Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Matt Kiely, Manager Medical Information, Abbott Vascular
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: AVD-640-0063
Record Dates: First submitted 2006-02-01; First posted 2006-02-07 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Carotid Artery Disease; Carotid Stenosis; Stroke; Atherosclerosis
Keywords: Carotid stenting; Carotid endarterectomy; Carotid artery disease with severe narrowing of the artery; Stroke prevention; cerebral infarction
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Stroke; Atherosclerosis; Cerebral Infarction | interventions — Methods

INTERVENTIONS:
Device: Carotid artery stenting with filter (interventional)

SUMMARY:
To collect clinical outcome and device performance data on the FDA 510(k)-cleared Emboshield® BareWire™ Rapid Exchange Embolic Protection System and FDA-approved Xact® Rapid Exchange Carotid Stent System when used under commercial use conditions by a broad group of physicians entering the study with differing carotid artery stenting experiences.

DETAILED DESCRIPTION:
This is a multi-center, observational, single arm, post-approval study enrolling the following study population:

* Subjects with neurological symptoms and >= 50% stenosis of the common or internal carotid artery by ultrasound or angiogram (visual estimate), or
* Subjects without neurological symptoms and >= 80% stenosis of the common or internal carotid artery by ultrasound or angiogram (visual estimate)
* The endpoint for the 1500 subjects enrolled will be a 30-day composite of death, stroke and myocardial infarction (MI).
* For the 500 subjects with 12 month follow-up, the endpoint will be a composite of stroke, death and MI at 30 days and ipsilateral stroke at 12 months (31-365 days).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who agree to participate in this study and have signed the IRB approved informed consent form.
* Subjects who are willing to have the Emboshield and/or the Xact inserted into the their vasculature.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The endpoint for the 1500 subjects enrolled will be a 30-day composite of death, stroke and myocardial infarction (MI).
For the 500 subjects with 12 month follow-up, the endpoint will be a composite of stroke, death and MI at 30 days and ipsilateral stroke at 12 months (31-365 days).

CONTACTS AND LOCATIONS:
Overall Officials: Don E Schwarten, MD, Study Chair — Abbott Medical Devices